CLINICAL TRIAL: NCT01753687
Title: Correlation of Different Signs for Assessment of Dry Eye Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: OPHT-300511
Record Dates: First submitted 2012-12-07; First posted 2012-12-20 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Dry Eye Syndrome
Keywords: break up time; tear film thickness; tear film osmolarity; objective scattering index; impression cytology; tear cytokines/chemokines; visual acuity; fluorescein staining
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 50 patients with dry eye syndrome (Other)
  Interventions: Other: Ocular scattering of the tear film; Other: Optical Coherence Tomography (OCT); Other: Measurement of tear film osmolarity

INTERVENTIONS:
Other: Ocular scattering of the tear film
  Other Names: OQAS, Visometrics, Spain
Other: Optical Coherence Tomography (OCT) — Tear film thickness as measured with OCT
Other: Measurement of tear film osmolarity
  Other Names: TearLab®, OcuSens Inc, San Diego, USA

SUMMARY:
Dry eye syndrome (DES) is a highly prevalent ocular condition inducing an inflammatory response of the ocular surface. Common symptoms include ocular discomfort, visual impairment and instability of the tear film with potential damage to the ocular surface.

The rationale of the present study is to compare signs as assessed with new methods such as measurement of tear film thickness, tear film osmolarity and scattering of the tear film with well established methods for assessment of the severity of DES (Break up time, staining of the cornea with fluorescein). Additionally, impression cytology and determination of tear cytokines/chemokines will be performed to obtain information about inflammatory processes on the ocular surface.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* History of dry eye syndrome for at least 3 months
* At least 2 symptoms of dry eye syndrome (foreign body sensation, burning, photophobia, blurred vision, pain, itching) and/or tear break up time < 10 seconds
* Normal ophthalmic findings except dry eye syndrome

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition that will interfere with the study aim as judged by the clinical investigator
* Wearing of contact lenses
* Intake of dietary supplements in the 3 months preceding the study
* Glaucoma
* Treatment with corticosteroids in the 4 weeks preceding the study
* Topical treatment with any ophthalmic drug in the 4 weeks preceding the study except topical lubricants
* Ocular infection or clinically significant inflammation
* Ocular surgery in the 3 months preceding the study
* Sjögren's syndrome
* Stevens-Johnson syndrome
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Break up time | once on the study day
  break up time of the tear film measured in seconds
Tear film thickness as measured with optical coherence tomography (OCT) | once on the study day
  tear film thickness measured in micrometers

SECONDARY OUTCOMES:
Visual Acuity | once on the study day
  Total number of letters read using ETDRS Charts
Tear film osmolarity | once on the study day
  Tear film osmolarity measured in mosmol/l
OSI (Objective Scattering Index) | once on the study day
  The objective scattering index will be measured using the OQAS system (Visiometrics, Spain)
Staining of the cornea with fluorescein | once on the study day
  The cornea will be divided into 5 regions (central, inferior, nasal, temporal, inferior) and each region will be graded from 0-4 in 0.5 steps as described in the Collaborative Longitudinal Evaluation of Keratoconus (CLEK) study.
Impression cytology | once on the study day
  After topical anesthesia of the eye, filter material is placed on the conjunctiva to obtain cytological samples, which will be prepared and evaluated.
Tear cytokines/chemokines | once on the study day
  Samples of 40 µl tears will be taken with a glass capillary and stored in vials. The concentrations of several cytokines and chemokines will be evaluated.
Subjective symptoms of dry eye syndrome | once on the study day
  a questionaire will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Schmidl D, Witkowska KJ, Kaya S, Baar C, Faatz H, Nepp J, Unterhuber A, Werkmeister RM, Garhofer G, Schmetterer L. The association between subjective and objective parameters for the assessment of dry-eye syndrome. Invest Ophthalmol Vis Sci. 2015 Feb 3;56(3):1467-72. doi: 10.1167/iovs.14-15814. PMID 25650419